CLINICAL TRIAL: NCT06935799
Title: Effectiveness of One-Minute Versus Two-Minute Cryoanalgesia in Nuss Surgery: A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of One-Minute Versus Two-Minute Cryoanalgesia in Nuss Surgery
Acronym: Cryo-One
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, Mateusz Ciopiński, Principal Investigator, Department of Pediatric Surgery and Organ Transplantation, CMHI, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37/KBE/2024
Record Dates: First submitted 2025-04-03; First posted 2025-04-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Pectus Excavatum; Funnel Chest
Keywords: cryoanalgesia; pain management; pectus excavatum; funnel chest
MeSH Terms: conditions — Funnel Chest; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One minute cryoanalgesia (Experimental)
  Interventions: Procedure: One minute intercostal nerves cryoanalgesia
- Two minutes cryoanalgesia (Active Comparator)
  Interventions: Procedure: Two minutes intercostal nerves cryoanalgesia

INTERVENTIONS:
Procedure: One minute intercostal nerves cryoanalgesia — One-minute cryoanalgesia will be applied bilaterally to each of the intercostal nerves from Th3 to Th7
  Arms: One minute cryoanalgesia
Procedure: Two minutes intercostal nerves cryoanalgesia — Two-minutes cryoanalgesia will be applied bilaterally to each of the intercostal nerves from Th3 to Th7
  Arms: Two minutes cryoanalgesia

SUMMARY:
Intercostal nerve cryoanalgesia has become a popular method for managing postoperative pain after Nuss procedure, showing greater effectiveness compared to epidural anesthesia and patient-controlled analgesia. However, the optimal duration of cryoanalgesia remains unknown. Most protocols use a two-minute cryoablation, although histological studies show similar changes with both one-minute and two-minute applications.

This is a pilot, single-center, randomized, double-blind study comparing the effectiveness of one-minute versus two-minute cryoanalgesia in treating pain in patients undergoing correction of pectus excavatum using the Nuss procedure. The aim of the project is to evaluate the validity of the research procedure and determine the sample size for the main study. Preliminary data on postoperative pain intensity, opioid consumption, duration of surgery, length of hospital stay, and complications will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pectus excavatum repair with MIRPE
* Written consent for corrective surgery with intraoperative cryoanalgesia
* Written consent to participate in the study
* Age >12 and < 18 years

Exclusion Criteria:

* History of previous thoracic surgeries
* Reoperation for chest deformity
* Contraindication for cryoanalgesia
* Presence of other conditions that may affect the course of the procedures and the assessment of their effectiveness and safety

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain level according to Numerical Rating Scale (NRS) | 1 week

SECONDARY OUTCOMES:
Opioid consumption | 1 week
Duration of the surgery | 1 day
Length of postoperative hospital stay | 1 week
Occurence of early complications | 30 days from the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Wybierz Województwo, Poland